CLINICAL TRIAL: NCT04917185
Title: Electro-acupuncture for Protracted Amphetamine Abstinence Syndrome : A Pragmatic Randomized Controlled Trial
Brief Title: EA for PAAS: A pRCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ren Yu-Lan, professor, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18ZDYF3417
Record Dates: First submitted 2021-05-26; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Substance Withdrawal Syndrome
MeSH Terms: conditions — Substance Withdrawal Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-Acupuncture group (Experimental): The patients in this group will be treated with electro-acupuncture for 30 minutes twice a week in a month. We conduct Nei Guan (PC6), Shen Men (HT7), ZuSanli (ST36), SanYinjiao (SP6) as the major points. Each time treating, according to other symptoms, we will give no more than 2 additional points.
  Interventions: Other: Electro-Acupuncture
- Wait-list group (No Intervention): We give no intervention to the patients this group during the whole experiment. When finishing, the same ways of treatment will be given to these patients.

INTERVENTIONS:
Other: Electro-Acupuncture — Acupuncture used for thousands years is part of traditional Chinese medicine. We use electro-acupuncture to treat our patients because it is more sufficient than traditional acupuncture and proved effectively treating protracted withdrawal syndrome of opioid use disorder. Paired alligator clips of the EA apparatus will be attached to the needle holders of Shenmen and Neiguan points on both sides. EA stimulation will last for 30 min with a continuous wave of 2/100Hz and intensity of 10-15 mA which patients can stand. All needles will be removed in 30 min and use a dry sterilised cotton ball to press the points in case of bleeding.
  Arms: Electro-Acupuncture group

SUMMARY:
In 2019, around 27 million people worldwide, corresponding to 0.5% of the adult population, have used amphetamine-type stimulants (ATS). More than one-third of these 27 million users of ATS were in East and South-East Asia. ATS are a group of synthetic psychostimulants including methamphetamine, amphetamine, 3,4-methylenedioxymethamphetamine (MDMA, ecstasy) and related substances. Although the biology underlying amphetamine withdrawal syndrome is not fully understood, amphetamine has been shown to produce long-lasting reductions in neuronal expression of dopamine neuronal markers. Abuse of these synthetic psychostimulants can lead to drug addiction, and subsequent withdrawal can cause a series of mental symptoms, such as anxiety, depression, confusion, insomnia, mood disturbances, cognitive impairments, and delusions. Some studies have shown two clear stages of ATS withdrawal syndrome: an acute phase lasting 7-10 days, and a subacute phase lasting a further 2 weeks or more, which is termed called "Protracted amphetamine abstinence syndrome (PAAS)".

The relevant literature has indicated that the majority of patients with ATS withdrawal disorders can experience depression, cognitive impairments, insomnia, and anxiety, especially during the PAAS stage. These symptoms may affect the treatment and finally lead to a relapse. Nowadays, pharmacological therapies are mostly symptom-targeted and show an ungratified effectiveness for amphetamine-type drugs. There is no a medication approved by Food and Drug Administration for use in the treatment of methamphetamine addiction. Therefore, the treatment of PAAS is essential for the treatment of ATS use disorders.

Traditional Chinese medicine (TCM), especially acupuncture, is effective in the treatment of withdrawal symptoms with few side effects. research on acupuncture detoxification originates from the treatment of opioid drug withdrawal. Studies have shown that acupuncture has high efficacy in the treatment of protracted abstinence symptoms after heroin addiction. This study hypothesizes that acupuncture has the same mechanism of action in the treatment of PAAS as in the treatment of protracted opioid abstinence syndrome. Therefore, investigators have designed a real-world-based pragmatic randomized controlled trial (pRCT) to determine the effectiveness of acupuncture in the treatment of PAAS and provide support for clinical decision-making.

Investigators conduct a pragmatic randomized controlled trials(pRCT) to observe the effect of acupuncture in a larger sample. It combines the advantages of randomization and real-world data, and the results can provide the best real-world evidence for the assessment of intervention effects or comparative effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients meet the diagnostic criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (21);
* A urine test for methamphetamine is negative.
* 18-60 years old, male or female, conscious, no aphasia, or mental retardation, primary school education or above, and able to understand the contents of the scales and cooperate with treatment;
* Did not participate in other clinical trials within 3 months;
* Signed the informed consent from.

Exclusion Criteria:

* Local trauma or infected persons who have received EA;
* Can' not tolerate EA, EA treatment, or allergic to EA needles;
* Pregnant or breastfeeding women;
* Serious disorders of the heart, liver, or kidney, or suicidal tendencies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Amphetamine Cessation Symptom Assessment | Change from baseline Amphetamine Cessation Symptom Assessment scores at 1 month.
  It consists of three subscales, namely, "anxiety and mood", "fatigue", and "craving". Items are scored on a five-point scale ranging from 0 to 4 with higher scores representing more severe Amphetamine Cessation Symptom

SECONDARY OUTCOMES:
Visual Analog Scale | Change from baseline Visual Analog Scale scores at 1 month.
  Determining the craving for amphetamine.The scores is from 0 to 10, and the higher scores means the more craving for amphetamine.
Hamilton Depression Scale | Change from baseline Hamilton Depression Scale scores at 1 month.
  Assessment for depression.And the interpretation of HAMD scores is as follows: <7, no depression; 7-17, mild depression; 17-24, moderate depression; and >24, severe depression.
Hamilton Anxiety Scale | Change from baseline Hamilton Anxiety Scale scores at 1 month.
  Assessment for anxiety. And the interpretation of HAMA scores is as follows: <7, no anxiety;7-14, mild anxiety; 14-20, moderate anxiety; 21-28, severe anxiety; and >29, extremely severe anxiety.
Pittsburgh Sleep Quality Index | Change from baseline Pittsburgh Sleep Quality Index scores at 1 month.
  The scores are from 0 to 21.Higher scores reflect worse sleep quality.
36-item Short Form Health Survey | Change from baseline 36-item Short Form Health Survey scores at 1 month.
  This questionnaire contains 9 parts: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health and Reported Health Transition.

CONTACTS AND LOCATIONS:
Overall Officials: Yulan Ren, PhD, Study Chair — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Affliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China